CLINICAL TRIAL: NCT04805008
Title: The Lactation Cookie Study
Brief Title: Lactation Cookie Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Ana M. Palacios, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 10036
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Breastfeeding
Keywords: Breastfeeding, lactation cookies, breast milk production
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will receive a generic bag of 57+/-1 grams of either lactation cookies or conventional cookies for 30 days.
  Investigators will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Lactation cookies
  Interventions: Other: Lactation cookies
- Control (Placebo Comparator): Control cookies
  Interventions: Other: Control cookies

INTERVENTIONS:
Other: Lactation cookies — 1 serving of 2 OZ of cookies per day for 30 consecutive days. These cookies will contain ingredients thought to increase breast milk production.
  Arms: Intervention
Other: Control cookies — 1 serving of 2 OZ of cookies per day for 30 consecutive days.
  The cookies will not contain ingredients thought to increase breast milk production.
  Arms: Control

SUMMARY:
Lactation cookies contain ingredients thought to increase breast milk production. Although these cookies are widely purchased and consumed with the intention to increase breast milk supply, no scientific investigation has explored the effects of lactation cookies on human breast milk production.

This study will evaluate the effects of a lactation cookie in breast milk production, relative to cookies without ingredients thought to increase breast milk production in exclusively breastfeeding mothers of healthy, term babies.

DETAILED DESCRIPTION:
Caring for an infant is demanding, and breastfeeding can become a stressful experience, particularly if mothers are concerned about their breast milk supply or whether their milk is nutritious enough to meet their infant's nutritional needs.

In the US, research suggests that about 60% of women perceive their breast milk as insufficient to meet their infant's nutritional needs. As a consequence, about one-fourth of women that perceive insufficient milk production wean their infants prematurely.

Lactation cookies contain ingredients thought to increase breast milk production and are widely consumed for this purpose. However, there is no research that has explored the effects of lactation cookies on breast milk supply. To answer this, the investigators plan a randomized controlled trial involving 176 exclusively breastfeeding mothers of 2-month-old infants. Participants will be randomized into "lactation cookies" or "control cookies" (cookies without ingredients thought to increase breast milk production" and will be asked to eat a bag (2 OZ) of cookies per day for 1 month.

ELIGIBILITY:
Inclusion Criteria

* Living in the contiguous continental 48 states in the US
* Mother of a healthy child born at 37 weeks or later from an uncomplicated birth
* Mother must be 18 years old or older
* Infant aged 2-months at enrollment
* Must intend to exclusively breastfeed infant for at least 3 months after birth
* Must have a working weight scale at home
* No formula use in 2 weeks prior to enrollment or plan to use during the study (1 month)
* Must not have any food or cookie ingredient allergies, dislikes, or contraindications to consume cookies
* Intending to bring the child to CDC recommended well-child visits

Exclusion Criteria

* Previous or current diagnosis of thyroid disease, epilepsy, psychosis, bipolar disorder
* Receiving treatment for depression or anxiety, or medications that may interfere with milk production (e.g. metoclopramide, chlorpromazine, domperidone, medroxyprogesterone, thyroid hormone).
* Substance use disorder
* Formula feeding or consuming other lactation boosting products during the study
* Having eaten lactation cookies in previous two weeks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Changes in breast milk production from baseline to 1-month post intervention | 1 month
  Assessed using the Roznowski 3-hour breast milk expression protocol (milk production hourly rate)

SECONDARY OUTCOMES:
Changes in perceived milk supply scores from baseline to 1-month post intervention | 1 month
  Assessed using the McCarter-Spaulding Perceived Insufficient Milk Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ana Palacios, MD, PhD, Principal Investigator — Indiana University, Bloomington; David Allison, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University - Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data related to the analysis and results of the primary and secondary outcomes listed herein will be available after deidentification.
Supporting Information: SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Palacios AM, Lemas DJ, Young BE, Parker E, Dickinson S, Marshall N, Sullivan KL, Wilt H, Cardel MI, Allison DB. Associations among Human Milk Polyunsaturated Fatty Acids and Infant Sleep Patterns: A Cross-Sectional Study. J Nutr. 2025 Oct;155(10):3426-3433. doi: 10.1016/j.tjnut.2025.07.021. Epub 2025 Aug 5. PMID 40754212
- [Derived] Palacios AM, Cardel MI, Parker E, Dickinson S, Houin VR, Young B, Allison DB. Effectiveness of lactation cookies on human milk production rates: a randomized controlled trial. Am J Clin Nutr. 2023 May;117(5):1035-1042. doi: 10.1016/j.ajcnut.2023.03.010. Epub 2023 Mar 14. PMID 36921902